CLINICAL TRIAL: NCT00370604
Title: Randomized Controlled Trial Examining the Effect of Small Versus Large Tuohy-type Epidural Needles on the Incidence and Severity of Postdural Puncture Headache
Brief Title: Effect of Small Versus Large Epidural Needles on Postdural Puncture Headache Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Canadian Anesthesiologists' Society (Other)
Responsible Party: Principal Investigator, Dr. Pamela Angle, Associate Professor, Director, Associate Scientist, Anesthesiologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1-PAngle
Record Dates: First submitted 2006-08-29; First posted 2006-08-31 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Post-Dural Puncture Headache
Keywords: Parturient; Obstetrics; Pregnancy; Labour; Labor; Headache; Epidural; Analgesia; Anesthesia; Anaesthesia
MeSH Terms: conditions — Post-Dural Puncture Headache; Headache; Agnosia | interventions — Catheters

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 19g needle, 23g catheter
  Interventions: Device: 19g Tuohy-type epidural needle, 23g catheter
- 2 (Active Comparator): traditional =>18g needle
  Interventions: Device: => 18g Tuohy-type needle

INTERVENTIONS:
Device: 19g Tuohy-type epidural needle, 23g catheter — Patients in the experimental group will receive a 23g 90cm adult length epidural catheter placed via a 19g Tuohy epidural needle (SIMS Portex, Hythe, UK). The 19g Tuohy needle is a standard 3½ inch length.
  Other Names: Health Canada Health Protection Branch (HPB) Licence # 6832; Smith's Medical epidural mini-kits 100/391/190
  Arms: 1
Device: => 18g Tuohy-type needle — Patients in the control arm will receive a traditional large gauge (16g, 17g or 18g Tuohy or Hustead) epidural needle and a traditional epidural catheter. Two control needles and two control catheters will be designated apriori by each institution for use in the study.
  Other Names: Hustead; Tuohy
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effect of 19g versus =>18g traditional Tuohy-type epidural needles on the incidence and severity of postdural puncture headache (PDPH).

DETAILED DESCRIPTION:
A headache is the most significant complication of dural puncture during epidural placement. This complication leads to longer hospital stays and many repeated visits to hospital for management. Women suffering from severe postdural puncture headache (PDPH) are often bedridden and unable to care for themselves or their babies.The efficacy of epidural blood patch as a "gold standard" therapy is over-estimated by the earlier, poor quality studies. The prevalence of dural puncture during epidural anesthesia using current techniques ranges from 0.03 to 6% in the literature. Of these patients, 70 to 80% will suffer from moderate to severe PDPH. Avoidance of dural puncture is always the goal. However, complete avoidance is unlikely using current techniques of needle placement. This study proposes another method of prevention (i.e., reducing the gauge of the epidural needles if it is shown to be suitable for continuous infusion in adults). Most of the risk factors for developing PDPH cannot be changed (e.g., younger age, female sex, low body mass index, history of migraines). However, epidural needle gauge is a modifiable risk factor. Evidence suggests that the use of smaller gauge epidural needles, like spinal needles, have the potential to reduce the incidence and severity of PDPH.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists status 1 to 2
* Must have provided written informed consent = or < 6cm cervical dilation
* Fetus 37 to 42 weeks gestation
* Must be able to read and write English well enough to provide written informed consent

Exclusion Criteria:

* BMI = or > 40
* Multiple gestation pregnancy
* Known contraindications to use of epidural analgesia
* Pregnancy-induced hypertension
* Investigator concern for maternal or neonatal welfare
* Receipt of spinal or epidural anesthesia within 14 days of labour epidural request
* Women with chronic headaches (defined as headaches that occur 15 or more days per month for more than 3 months)
* Already participated in study
* History of narcotic abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1081 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Incidence of postdural puncture headache | within the first 14 days of epidural placement

SECONDARY OUTCOMES:
PDPH characteristics (quality, distribution, postural versus non-postural nature, associated symptoms) | within first 14 days post-epidural placement, and if necessary, up to 1 year post-epidural placement
Severity of pain related to PDPH | within first 14 days post-epidural placement, and if necessary, up to 1 year post-epidural placement
Degree of dysfunction and disability related to PDPH symptoms | within first 14 days post-epidural placement, and if necessary, up to 1 year post-epidural placement
Duration of PDPH-related symptoms | within first 14 days post-epidural placement, and if necessary, up to 1 year post-epidural placement
Pain and pain relief (first and second stage labor analgesia following epidural placement and overall pain relief) as rated by the patient, compared between groups | within 24 hours of epidural placement
Incidence of persistent PDPH symptoms between groups | at 6 weeks post-epidural placement
Number and timing of epidural blood patches received, total number of epidural blood patches received until symptom resolution | within the first 6 weeks of epidural placement
Risk of delayed block failure for continuous labour analgesia in patients receiving a 19g Tuohy epidural needle and 23g catheter | after first 30 minutes of successful initiation (requiring epidural reinsertion)
Risk of requiring use of an alternative method of anesthesia for operative delivery in patients receiving successful epidural initiation with a 19g Tuohy epidural needle and a 23g catheter | during labour and delivery
Incidence of significant adverse events in each group | up to 1 year post-epidural placement
Patient ratings of overall pain relief compared between groups | during labour and delivery
Anesthesiologist satisfaction with the 19g Tuohy epidural needle and 23g catheter compared with traditional Tuohy type epidural needles and traditional catheters | during labour and delivery

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J Angle, MD, MSc, Principal Investigator — Women's College Hospital at Sunnybrook Health Sciences Centre
Locations (4):
- Canada (4):
  - British Columbia Women's Hospital and Health Centre, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - St. Joseph's Hospital, London, Ontario
  - Sunnybrook Health Sciences Centre at Women's College Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Angle PJ, Hussain K, Morgan A, Halpern SH, Van der Vyver M, Yee J, Kiss A. High quality labour analgesia using small gauge epidural needles and catheters. Can J Anaesth. 2006 Mar;53(3):263-7. doi: 10.1007/BF03022213. PMID 16527791